CLINICAL TRIAL: NCT03370276
Title: A Phase I/II Study of Concurrent Cetuximab and Nivolumab in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Cetuximab & Nivolumab in Patients With Recurrent/Metastatic Head & Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other); Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19178
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx; Squamous Cell Carcinoma of the Larynx; Squamous Cell Carcinoma of the Oral Cavity; Squamous Cell Carcinoma of the Hypopharynx; Squamous Cell Carcinoma of the Paranasal Sinus; Head and Neck Squamous Cell Carcinoma; Squamous Cell Cancer; Head and Neck Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms, Squamous Cell | interventions — Nivolumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase I - Affiliate Sites Only (Experimental): Nivolumab and dose escalation of Cetuximab.
  Dose Level 1:
  Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 500 mg/m^2; Nivolumab 240 mg.
  Dose Level -1:
  Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 250 mg/m^2; Nivolumab 240 mg.
  Interventions: Drug: Nivolumab; Drug: Cetuximab
- Phase I - Moffitt Site Only (Experimental): Nivolumab and dose escalation of Cetuximab.
  Dose Level 1:
  Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 500 mg/m^2; Nivolumab 240 mg.
  Dose Level -1:
  Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 250 mg/m^2; Nivolumab 240 mg.
  Interventions: Drug: Nivolumab; Drug: Cetuximab
- Phase II - Affiliate Sites Only (Experimental): Nivolumab and Cetuximab at recommended Phase II dose (RP2D).
  Interventions: Drug: Nivolumab; Drug: Cetuximab
- Phase II - Moffitt Site Only (Experimental): Nivolumab and Cetuximab at recommended Phase II dose (RP2D).
  Interventions: Drug: Nivolumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms.
  Other Names: Opdivo
Drug: Cetuximab — Cetuximab intravenously (IV) at 500 mg/m^2 or 250 mg/m^2 as outlined in the treatment arms.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to find out if the combination of two established anti-cancer therapies are beneficial in participants with Head and Neck Squamous Cell Carcinoma (HNSCC). Specifically, investigators want to determine if the combination of Cetuximab and nivolumab can help people with advanced cases of HNSCC. Both cetuximab and nivolumab have been used separately to treat HNSCC and are Food and Drug Administration (FDA) approved in this type of cancer.

DETAILED DESCRIPTION:
PHASE I: Participants will be enrolled sequentially and treated at Dose Level 1, or Dose Level -1, every 2 weeks for 12 cycles or until discontinuation.

Each cycle is 4 weeks. Cetuximab is given alone in lead-in period at Day -14 before Cycle 1 only. In all subsequent doses starting Cycle 1 Day 1, nivolumab and cetuximab will be given concurrently. Dose limiting toxicity (DLT) assessment will be performed during Cycle 1 and will start with the initiation of the combination of cetuximab and nivolumab (4 weeks).

PHASE II: Once the maximum tolerated dose (MTD) or the recommended phase II dose of cetuximab is determined in Phase I, accrual to the phase II will begin.

FOLLOW-UP: Participants will be followed for 2 years from End of Treatment. The imaging studies will be performed every 8 weeks (2 cycles) of the treatments during Cycle 1-6 and then every 12 weeks during Cycle 7-12 as per standard of care. Patient will be followed by treating physicians as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed squamous cell carcinoma of oral cavity, oropharynx, paranasal sinuses, nasal cavity, hypopharynx, or larynx. Squamous cell carcinoma of unknown primary in cervical lymph node can be included only if p16 status is positive.
* Must have recurrent or metastatic HNSCC stage III/IV that is not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).Patients with persistent disease following radiation therapy administered with a chemotherapy sensitizer may also be included.
* Must have progressed on at least one prior line of chemotherapy, targeted therapy, palliative radiation, and/or biological therapy regimen for their recurrent and/or metastatic HNSCC. However, if patients are likely to be intolerant to standard first-line systemic chemotherapy, the patients are eligible to enroll to this study as the first-line therapy. Additionally, patients with persistent disease or platinum-refractory recurrent disease may enroll in this study as a first-line therapy.
* Must NOT have any systemic therapy for recurrent and/or metastatic disease except if given as a part of a multimodality treatment (i.e. re-irradiation and systemic therapy for curable intent of locally recurrent disease).
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as outlined in RECIST version 1.1.
* Must be ≥ 18 years of age.
* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Must have normal organ function: Absolute neutrophil count > 1,500/μL; Hemoglobin > 9 g/dL; Platelets > 100,000/μL; Total bilirubin ≤ 1.5 mg/dL X institutional upper limits of normal (ULN); AST (SGOT)/ALT (SGPT) < 3 X institutional ULN (or 5.0 X the ULN in the setting of liver metastasis); Serum creatinine of ≤ 1.5 X ULN or creatinine clearance > 40 mL/minute (using Cockcroft/Gault formula): Female creatinine clearance = (140 - age in years) x weight in kg x 0.8572 x serum creatinine in mg/ dL; Male creatinine clearance = (140 - age in years) x weight in kg x 1.0072 x serum creatinine in mg/dL.
* Participants, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods). Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Have experienced grade 3 or above skin toxicity from prior Epidermal growth factor receptor (EGFR) inhibiting therapy.
* Have experienced grade 3 or above toxicity from prior anti-PD1 therapy.
* Have p16 negative squamous cell carcinoma of unknown primary in cervical lymph node.
* Patients with primary nasopharynx or salivary gland cancers.
* Patients who have had chemotherapy, biological therapy or definitive radiation within 4 weeks of the study enrollment or those who have not recovered from adverse events to ≤ Grade 1 due to agents administered more than 4 weeks earlier.
* Had undergone any major surgery within 4 weeks of study enrollment.
* Had undergone any palliative radiation within 2 weeks of study enrollment.
* Have had other investigational agents within 4 weeks or 5 half-lives, whichever is shorter, of the study enrollment.
* Have known leptomeningeal metastases or untreated or symptomatic brain metastases. Treated, asymptomatic brain metastasis can be included.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune disease requiring systemic steroids, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Have clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency.
* Have uncontrolled or poorly controlled hypertension (>180 mmHg systolic or > 130 mmHg diastolic) at the time of enrollment.
* Prior treatment with a combination of cetuximab and a PD-1/PD-L1 inhibitor. Prior treatment with cetuximab or a PD-1/PD-L1 inhibitor is allowed as long as not previously given in combination.
* A history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab and/or nivolumab.
* Pregnant or breast-feeding.
* Known active HIV, Hep B, or Hep C infection. If not clinically indicated, the patients do not need to be tested.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine H. Chung, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - The Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Wang X, Muzaffar J, Kirtane K, Song F, Johnson M, Schell MJ, Li J, Yoder SJ, Conejo-Garcia JR, Guevara-Patino JA, Bonomi M, Bhateja P, Rocco JW, Steuer CE, Saba NF, Chung CH. T cell repertoire in peripheral blood as a potential biomarker for predicting response to concurrent cetuximab and nivolumab in head and neck squamous cell carcinoma. J Immunother Cancer. 2022 Jun;10(6):e004512. doi: 10.1136/jitc-2022-004512. PMID 35676062
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in lead-in were included in Cohort A for outcome measure data.
Groups:
- Phase I - Lead in: Nivolumab and dose escalation of Cetuximab.
  Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 500 mg/m^2; Nivolumab 240 mg.
  Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms.
  Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2.
- Phase II- Cohort A: Patients who had progressed on at least one prior line of treatment for their recurrent and/or metastatic HNSCC
  Participants were treated with Nivolumab and Cetuximab at recommended Phase II dose (RP2D). Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms. Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2.
- Phase II - Cohort B: Patients who have not had any prior treatment for their recurrent and/or metastatic HNSCC
  Participants were treated with Nivolumab and Cetuximab at recommended Phase II dose (RP2D). Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms. Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2.
Period: Overall Study
Arm/Group | Phase I - Lead in | Phase II- Cohort A | Phase II - Cohort B
Started | 3 | 44 | 48
Completed | 3 | 42 | 43
Not Completed | 0 | 2 | 5
Not completed — Death | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Phase I - Lead in: Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 500 mg/m^2; Nivolumab 240 mg.
  Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms.
- Phase II - Cohort A: Patients who had progressed on at least one prior line of treatment for their recurrent and/or metastatic HNSCC
  Participants were treated with Nivolumab and Cetuximab at recommended Phase II dose (RP2D). Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms. Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2 or 250 mg/m^2 as outlined in the treatment arms.
- Phase II - Cohort B: Patients who have not had any prior treatment for their recurrent and/or metastatic HNSCC
  Participants were treated with Nivolumab and Cetuximab at recommended Phase II dose (RP2D). Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms. Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2 or 250 mg/m^2 as outlined in the treatment arms.
- Total: Total of all reporting groups
Arm/Group | Phase I - Lead in | Phase II - Cohort A | Phase II - Cohort B | Total
Number analyzed (Participants) | 3 | 44 | 48 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 24 | 32 | 58
  >=65 years | 1 | 20 | 16 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 15 | 23
  Male | 2 | 37 | 33 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 41 | 45 | 89
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 3 | 6
  White | 3 | 39 | 42 | 84
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 44 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose
Description: Maximum Tolerated Dose (MTD).. The target Dose Limiting Toxicity (DLT) rate is <25%. The MTD will be defined as the dose of cetuximab and nivolumab in which <1 of 3 patients experience a DLT or <2 of 6 patients experience a DLT with the next higher dose having at least 2 patients experiencing a DLT. The MTD is the highest dose at which at most 1 of 6 patients has a DLT. This study will utilize the Cancer Therapy Evaluation Program CTCAE version 4.1 for toxicity and event reporting. Dose-limiting toxicities will be observed until patients have completed Cycle 1 (4 weeks).
Time Frame: Up to 12 months
Measure: Number; unit: mg/m^2
Groups:
- Phase I - Lead in: Nivolumab and dose lead in of Cetuximab.
  Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 500 mg/m^2; Nivolumab 240 mg.
  Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms.
  Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2 or 250 mg/m^2 as outlined in the treatment arms.
Arm/Group | Phase I - Lead in
Number analyzed (Participants) | 3
mg/m^2 | 500

2. Primary Outcome: Phase II: Overall Survival (OS)
Description: One year overall survival of concurrent cetuximab and nivolumab in patients with recurrent and/or metastatic HNSCC. OS: The length of time from the start of treatment until death by any cause.
Time Frame: Up to 24 months
Population: Evaluable participants
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Phase I Lead in + Phase II: Cohort A: Patients who had progressed on at least one prior line of treatment for their recurrent and/or metastatic HNSCC
  Participants were treated with Nivolumab and Cetuximab at recommended Phase II dose (RP2D). Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms. Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2 or 250 mg/m^2 as outlined in the treatment arms.
Arm/Group | Phase I Lead in + Phase II: Cohort A | Phase II - Cohort B
Number analyzed (Participants) | 45 | 43
months | 11.4 [9.4 to 14.4] | 20.2 [15.7 to 24.7]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Complete Response (CR): The disappearance of all measurable lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameters of measureable lesions, taking as reference the baseline sum longest diameter. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s). Stable Disease (SD): Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease. To be assigned a status of stable disease, measurements must have met the stable disease criteria at least once after study entry at a minimum interval of 6 weeks.
Time Frame: Up to 48 months
Population: Participants evaluable for response
Measure: Number; unit: percentage of participants responded
Arm/Group | Phase I Lead in + Phase II: Cohort A | Phase II - Cohort B
Number analyzed (Participants) | 43 | 42
percentage of participants responded | 22 | 37

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progressive Disease (PD): At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).
Time Frame: at 12 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Lead in + Phase II: Cohort A | Phase II - Cohort B
Number analyzed (Participants) | 45 | 43
months | 3.35 [2.56 to 7.13] | 6.15 [3.06 to NA] — Not reached

5. Secondary Outcome: Number of Study Treatment Related Adverse Events
Description: Related adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) V4.1. An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product.
  A serious adverse event (SAE) is defined as any AE that results in death, is immediately life-threatening, results in persistent or significant disability/incapacity, requires or prolongs patient hospitalization, is a congenital anomaly/birth defect, or is to be deemed serious for any other reason if it is an important medical event when based on appropriate medical judgement that may jeopardize the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.
Time Frame: Up to 48 months
Population: Evaluable participants
Measure: Number; unit: events
Arm/Group | Phase I Lead in + Phase II: Cohort A | Phase II - Cohort B
Number analyzed (Participants) | 45 | 43
events
  Grade 1 | 115 | 228
  Grade 2 | 105 | 142
  Grade 3 | 23 | 27
  Grade 4 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events collected from on study date to 30 days after completion of study therapy, approximately 2 years. All participants were followed for events, whether or not evaluable.
Groups:
- Phase I - Lead in: Nivolumab and dose escalation of Cetuximab.
  Lead-in Day -14 before Cycle 1 only: Cetuximab 500 mg/m^2; Nivolumab - none. Cycle 1 Day 1 and all subsequent doses every 2 weeks (Q2W): Cetuximab 500 mg/m^2; Nivolumab 240 mg.
  Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms.
  Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2 or 250 mg/m^2 as outlined in the treatment arms.
- Phase II- Cohort A: Patients who had progressed on at least one prior line of treatment for their recurrent and/or metastatic HNSCC
  Participants were treated with Nivolumab and Cetuximab at recommended Phase II dose (RP2D). Nivolumab: Nivolumab intravenously (IV) at 240 mg as outlined in the treatment arms. Cetuximab: Cetuximab intravenously (IV) at 500 mg/m^2 or 250 mg/m^2 as outlined in the treatment arms.
Arm/Group | Phase I - Lead in | Phase II- Cohort A | Phase II - Cohort B
All-Cause Mortality (participants affected / at risk) | 2/3 | 35/44 | 33/48
Serious Adverse Events (participants affected / at risk) | 3/3 | 19/44 | 19/48
Other Adverse Events (participants affected / at risk) | 3/3 | 43/44 | 45/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Lead in (N=3) | Phase II- Cohort A (N=44) | Phase II - Cohort B (N=48)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Renal and urinary disorders -Other (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1)
Death, NOS (General disorders) | 0 (0) | 2 (2) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — PEG tube re-placement
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Neoplasms benign, malignant and unspecified-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6) | 3 (3) — Disease progression
Atrial fibrilation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 7 (11)
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Bacterial pneumonia
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Parasthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Anemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications -Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Feeding tube displaced by patient
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Intra-abdominal infection
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — PEG tube malfunction/redness
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 1 (1) | 0 (0) — G tube dysfunction
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Duodenitis
Sudden death, NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — tracheostomy obstruction by mucous
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Lead in (N=3) | Phase II- Cohort A (N=44) | Phase II - Cohort B (N=48)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 5 (6) | 4 (5)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 7 (11)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (6) | 7 (13)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 5 (6) | 14 (47)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 8 (8) | 9 (10)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (5) | 5 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 11 (20)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (3)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Blurred vision (Eye disorders) | 0 (0) | 2 (3) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (4)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 16 (17) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 6 (7)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 8 (16) | 12 (22)
Dizziness (Nervous system disorders) | 1 (2) | 5 (5) | 7 (11)
Cardiac disorders - Other (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 9 (11)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (10) | 23 (28)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (5) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (13) | 9 (19)
Ear and labyrinth disorders -Other (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (4)
Edema face (General disorders) | 0 (0) | 4 (5) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 5 (6) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders -Other (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 3 (3) | 5 (7)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 12 (15) | 6 (9)
Fatigue (General disorders) | 2 (4) | 17 (29) | 15 (28)
Fever (General disorders) | 0 (0) | 3 (3) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 10 (11) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (2) | 6 (11)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 5 (5) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (3)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 7 (8) | 5 (6)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 5 (7) | 11 (54)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 8 (15) | 8 (81)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (10) | 5 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 11 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 8 (16) | 16 (49)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 5 (10) | 8 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 7 (14) | 14 (29)
Hypotension (Vascular disorders) | 0 (0) | 3 (4) | 4 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 6 (6) | 7 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 6 (11) | 6 (11)
Infusion related reaction (General disorders) | 1 (2) | 1 (1) | 9 (13)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5) | 8 (9)
Intraoperative renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 2 (2) | 5 (5)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1) | 6 (6)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 3 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 6 (8) | 11 (34)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 3 (5) | 6 (10)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 5 (7) | 7 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 4 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 9 (10)
Nausea (Gastrointestinal disorders) | 1 (2) | 9 (13) | 11 (18)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 4 (4)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 8 (8) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (7) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 7 (7) | 9 (25)
Paresthesia (Nervous system disorders) | 0 (0) | 3 (3) | 6 (7)
Paronychia (Infections and infestations) | 0 (0) | 7 (11) | 12 (30)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 2 (3)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (8) | 10 (13)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5) | 21 (36) | 31 (63)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 4 (10)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 9 (15)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (3) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (15) | 19 (34)
Skin infection (Infections and infestations) | 1 (1) | 3 (4) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 4 (4)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4)
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 5 (6)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (6)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (7) | 7 (20)
Weight gain (Investigations) | 0 (0) | 0 (0) | 4 (11)
Weight loss (Investigations) | 0 (0) | 7 (9) | 8 (15)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 4 (8)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The rights to publish the results of the study are vested in Moffitt. Subsite is free to publish any academic article, presentation or abstracts of the study results (including supporting data) twelve months after the conclusion or termination of the study provided that any such manuscript is first submitted to Moffitt sixty days prior to the proposed publication date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03370276/Prot_SAP_000.pdf